CLINICAL TRIAL: NCT03801096
Title: Project RAD: A Brief Intervention for Young Adult Alcohol or Marijuana Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Marcel de Dios, PhD, Assistant Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00001218
Record Dates: First submitted 2019-01-08; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Alcohol; Use, Problem; Marijuana Usage
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Two-group randomized controlled trial (RCT) design
Who Masked: Outcomes Assessor
Masking Description: Research Assistant collecting data will be blinded to condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrative Based Therapuetic Assessment (Experimental)
  Interventions: Behavioral: Narrative Based Therapuetic Assessment (NbTa)
- Health Education (HE) (Active Comparator)
  Interventions: Behavioral: Health Education Control Condition (HE)

INTERVENTIONS:
Behavioral: Narrative Based Therapuetic Assessment (NbTa) — The NbTa interventiom will guide participants through an exploration of their human experience through stories and narratives. The interventionist will facilitate a collaborative process by which participants will explore the unique themes and meanings of their personal narrative (Parry & Doan, 1994) with respect to alcohol and drug use. In addition, participants will also be guided towards considering the re-authorship of personal narratives. The techniques utilized in NbTa aim to dislodge problem saturated narratives and derive more complete personal narratives and meanings (White & Epston, 1990).
  Arms: Narrative Based Therapuetic Assessment
Behavioral: Health Education Control Condition (HE) — The Health Education session is a didactic 45-minute session that focusses on three health-related topics: 1) Sleep, 2) Physical Activity, and 3) Nutrition. The goal of the session is to present health-related information to participants through videos and dydadic presentation.
  Arms: Health Education (HE)

SUMMARY:
This is a pilot study of the feasibility, acceptability, and effectiveness of a brief, one-session intervention for a diverse sample of 44 young adults who report alcohol binge drinking or marijuana use in the past month. The proposed study will utilize a two-group randomized controlled trial (RCT) design. Participants will be randomized to one of two interventions conditions: 1) Narrative-based Therapeutic Assessment (NbTa) or 2) Health Education (HE) control condition. Participants will be assessed on their 7- and 30-day alcohol and marijuana use at baseline and at 6 month follow-up.

DETAILED DESCRIPTION:
This study is a preliminary examination of the feasibility, acceptability, and effectiveness of a brief, one-session intervention for a diverse sample of young adults who report alcohol binge drinking or marijuana use in the past month. The proposed study will utilize a two-group pilot randomized controlled trial (RCT) design. Participants will be randomized to one of two interventions conditions in a 1:1 distribution using a standard urn randomization technique stratified by gender and substances used in the past month only, alcohol AND marijuana). Participants will be randomized to either: 1) Narrative- based Therapeutic Assessment (NbTa) or 2) Health Education (HE) control condition.

10.2 Recruiment Potential participants will be recruited using an IRB approved flyer posted at locations in the greater Houston area that are likely to be frequented by our target young adult population (e.g. college campuses, gyms, coffee shops, grocery stores, etc). Potential participants will also be recruited through online advertising, as well as through email and social media advertisements. Individuals that are interested in participating in the study will call the study phone number. Participants will also have the opportunity to contact the study via a secure email address.

Upon arrival at the study site, the RA will greet the participant and begin the Informed Consent Process. The RA will provide the participant with a verbal and written overview of the study including aims, risks, compensations, and all study procedures. The RA will provide each potential participant with the opportunity to ask questions about the study. The RA will emphasize the voluntary nature of the study and tell participants that they may withdraw at any time during the study. Potential participants will be given as much time as needed to review the written (Informed Consent Document [ICD]) and will be given a copy for their records. The ICD will include the contact information of the PI as well as the UH IRB. Participants that agree to participate will sign the ICD and the RA will document the entire process. After Informed Consent has been obtained, the participant will be rescreened in order to verify that participants continue to meet inclusion and exclusion criteria.

Once eligibility has been re-established the RA will provide participants with a computer tablet that participants will be instructed to use to complete the study questionnaires. The questionnaires will be administered using Qualtrics and the data will be stored on a secure server with firewall and password protection maintained by the College of Education's Center for Information Technology in Education. While the participant completes the questionnaires on the tablet the RA will be available for questions or concerns. Participants will be instructed to complete the questionnaire to the best of their ability. Participants will also be told that if they do not feel comfortable with any questions, they may skip them. Participants will be offered bottled water and will be able to take bathroom breaks as needed during the assessment. A full list of measures is provided in Appendix 2 with the timepoint to be given. The Investigative team has conducted two pilot mock completions of the assessment battery and it takes approximately 1 to 1.5 hours to complete the baseline assessment and 30-45 minutes to complete the follow-up assessment. After completing the questionnaires, participants will complete two biological tests to confirm their self-reported substance use. First, participants will be asked to provide a urine sample. The RA will provide the participant with a collection cup and instructions for the participant to collect the sample. Participants will not be directly observed while providing the urine sample. The RA will wait outside of the bathroom with an nondescript collection bin. The urine sample cup is equipped with built-in tests for the thirteen most common substances used including alcohol, marijuana, and other drugs. The test cup will indicate a positive or negative result for each substance tested and the RA will document the result and discard the collection cup. The sealed cup containing the urine sample can be discarded in the restroom and is not considered a biohazard. It will not contain any identifying information on it and the test strips become unreadable within 20 minutes. Once the urine sample results are documented, the RA will collect a sample of expired carbon monoxide using a Bedfont Micro+ Smokerlyzer®. This test measures the level of carbon monoxide, which is an indicator of combustible smoking including marijuana and tobacco use. The collection of this sample will involve participants taking a deep breath, holding it for 15 seconds, and exhaling into a handheld electronic device. The report will range from 0-500ppm, and the sensor is accurate by 1ppm. The RA will document the results on a CO test results form.

After the two biological tests have been completed, the RA will schedule the participant's 6-month follow-up visit. The RA will remind participants about the expected duration of the 6 month Follow-Up Visit.

Intervention The RA will then escort the participant to the interventionist's office and will introduce the participant and the interventionist to one another. Once the RA has left, the interventionist will open the presequenced randomization envelope and document the participant's study group. The interventionist will inform the participant of the group they have been randomized to. Participants randomized to the NbTa intervention condition will receive a 45-minute Narrative-Based Therapeutic Assessment intervention session. Those randomized to the Health Education control condition will receive a time-matched intervention session that will involve the viewing of health-related educational videos with a brief discussion. The investigative team has used the Health Education Intervention as a control group intervention in a previous trial of substance users (de Dios, Cano, Vaughan, Childress, McNeel, & Niaura, Under Review). All NbTa sessions will be audio/video recorded and this data will be stored on a secure password protected institutional server. The Health Education sessions will not be audio/video recorded. Participants may choose not to be audio/video recorded for any reason. The recordings are not a condition of participation. For the delivery of both interventions, manuals will be used to ensure standardization of intervention delivery as well as provide a basis for evaluating interventionist adherence.

Upon completing the intervention session, participants will complete the SSSE to rate their satisfaction with the content of the session.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 25.
* Able to speak and read the English language.
* Agree to participate in the study and be available for two study visits that will occur at baseline and approximately 6-month after the baseline visit.
* Report at least 1 alcohol binge drinking episode in the past month (binge drinking is defined as 4 or more drinks in a 2 hour period for women, 5 or more drinks in a 2 hour period for men (NIAAA, 2004) OR report the use of marijuana on at least 1 occasion in the past month.
* Have access to an email account or phone number to communicate with study personnel.
* Identify as a member of a minority group, disadvantaged group, or marginalized based on race, ethnicity, heritage, immigration status, gender, sexual orientation, religion, and disability status.

Exclusion Criteria:

* In the past month, consumed an average of 7 or more drinks per week for females or 14 or more drinks per week for males.
* Marijuana use on 4 or more days per week in the past month.
* A pattern of impaired functioning due to alcohol or marijuana use during the past month;
* In the past year, family members, close friends, or medical providers have expressed concerns about their alcohol or marijuana use and have advised them to quit.
* A history of a Substance Use Disorders (Alcohol; Amphetamines; Cannabis; Cocaine; Hallucinogens; Opioids; Phencyclidine; and Sedatives, Hypnotics and Anxiolytics).
* A history of a chronic and/or severe psychiatric disorder that would interfere with participation (i.e., Schizophrenia, Delusional Disorder, Schizoaffective Disorder, Bipolar Disorder, or a Mood Disorder with Psychotic Features).
* Unavailable for a 2.5 hour baseline visit and a follow-up visit 6 months post baseline.
* Unable to provide contact information to allow for study related communication.
* Pregnant or nursing.
* Identified as a UH student that the PI (Dr. Marcel de Dios) has had or will likely have direct access to or influence over through academic activities such as coursework, advising, or research mentoring.
* Identified by the study PI as unsuitable for participating in the study due to significant circumstances that would interfere with participation including threatening behavior or an inability/unwillingness to respond to basic study related questions and instructions.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All self-represented gender identities will be included.
Enrollment: 44 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Weekly Alcohol Use Frequency at 6 month follow-up | 6 months after baseline
  Self-reported days of alcohol use in the past 7 days captured and computed using the Timeline Follow Back (Sobel & Sobel, 1992).
Monthly Alcohol Use Frequency at 6 month follow-up | 6 months after baseline
  Self-reported days of alcohol use in the past 30 days captured and computed using the Timeline Follow Back (Sobel & Sobel, 1992).
Weekly Marijuana Use Frequency at 6 month follow-up | 6 months after baseline
  Self-reported days of marijuana use in the past 7 days captured and computed using the Timeline Follow Back (Sobel & Sobel, 1992) and confirmed with Urine drug screening tests.
Monthly Marijuana Use Frequency at 6 month follow-up | 6 months after baseline
  Self-reported days of marijuana use in the past 30 days captured and computed using the Timeline Follow Back (Sobel & Sobel, 1992) and confirmed with Urine drug screening tests.

IPD SHARING:
Plan to Share IPD: No